CLINICAL TRIAL: NCT01017536
Title: Phase II Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of AERAS-402 in HIV-infected, BCG-vaccinated Adults With CD4+ Lymphocyte Counts Greater Than 350 Cells/mm3
Brief Title: Safety and Immunogenicity of AERAS-402 in HIV-infected, Bacillus Calmette-Guerin (BCG)-Vaccinated Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-017-402
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-07

CONDITIONS: Tuberculosis; HIV Infections
Keywords: HIV; Tuberculosis; Vaccine
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — AERAS-402

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Thirteen subjects received placebo vaccine that did not contain any AERAS-402.
  Interventions: Biological: Placebo
- Investigational Vaccine (Experimental): Thirteen subjects received active vaccine 3 x 10^10 vp AERAS-402.
  Interventions: Biological: AERAS-402

INTERVENTIONS:
Biological: AERAS-402 — AERAS-402 is a replication-deficient serotype 35 adenovirus containing DNA that expresses a fusion protein of three Mycobacterium tuberculosis (Mtb) antigens: 85A, 85B and TB10.4.
  Arms: Investigational Vaccine
Biological: Placebo — Placebo was the identical buffer solution in which AERAS-402 is formulated.
  Arms: Placebo

SUMMARY:
This was a Phase II, randomized, double-blind, placebo-controlled trial conducted at 1 site in South Africa. A total of 26 subjects were randomized 1:1 to receive 2 doses of either AERAS-402 at 3 x 10^10 vp (N=13) or placebo (N=13) on Study Days 0 and 28. Dose-escalation to a second group of 40 subjects was planned, but although no safety concerns were identified, the sponsor decided not to continue the study.

DETAILED DESCRIPTION:
Further study details as provided by Aeras.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years through 45 years (i.e., subject had not yet reached his/her 46th birthday at day of randomization).
2. Had completed the written informed consent process prior to undergoing any screening evaluations.
3. Had BCG vaccination at least 5 years previously, documented by medical history or presence of scar.
4. Females: Ability to avoid pregnancy for at least 6 months after receiving the last study vaccination: Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) must have avoided pregnancy from 28 days prior to administration of the study vaccine and must have agreed to avoid pregnancy through at least 6 months after receiving the last study vaccination. Acceptable methods of avoiding pregnancy included a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), or use of a combination of at least two forms of acceptable contraception: hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), and the use of a condom or a diaphragm; or the use of a condom or a diaphragm combined with spermicide.
5. Was able to carry out activities of daily living independently.
6. Had Body Mass Index (BMI) of at least 19 (wt./ht.2) by nomogram.
7. Had ability to complete follow-up period as required by the protocol.
8. Was able and willing to commit to avoiding elective surgery for at least 6 months after receiving the last study vaccination.
9. Was able and willing to stay in contact with the study site for the duration of the study.
10. Had committed to simultaneous enrollment in Aeras Vaccine Development Registry Protocol.
11. Had laboratory evidence of human immunodeficiency virus (HIV) infection, defined as a positive HIV-1 ELISA test plus a positive confirmatory test (e.g., a second HIV-1 ELISA, PCR, or rapid ELISA).
12. Had four (4) (for Group 1) or three (3) (for Group 2)* CD4+ lymphocyte count tests, each performed at least four days apart within the 42-day screening period, with at least three (for Group 1) or two (for Group 2) CD4+ lymphocyte count results greater than 350 cells / mm3.
13. Not currently receiving antiretroviral drugs.
14. Committed to not participate in any other clinical trials during the first 12 months of participation in this study.

Exclusion Criteria:

1. Acute illness.
2. Fever ≥37.5°C.
3. Significant symptomatic infection.
4. Used immunosuppressive medication within 42 days prior to randomization (inhaled and topical corticosteroids were permitted).
5. Received immunoglobulin or blood products within 42 days prior to randomization.
6. Received any investigational drug therapy or vaccine within 182 days prior to randomization.
7. History of having received any adenovirus-vector-based vaccine.
8. Medical history that may have compromised the evaluation of safety of the subject in the study (e.g., diabetes, seizure disorder, sickle cell disease).
9. Pregnant or breastfeeding female, or intention to become pregnant during the study within 6 months after receiving the last study vaccination.
10. Liver function tests >Grade 2 per the toxicity table.
11. Currently receiving treatment for TB, or evidence of active TB disease based on history, physical examination, chest X-ray, or laboratory evaluation (INH prophylaxis was permitted).

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, MD, PhD, Principal Investigator — Aurum Institute; Bernard Landry, MPH, Study Director — Aeras
Locations (1):
- Aurum Institute, Klerksdorp, North West, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Churchyard GJ, Snowden MA, Hokey D, Dheenadhayalan V, McClain JB, Douoguih M, Pau MG, Sadoff J, Landry B. The safety and immunogenicity of an adenovirus type 35-vectored TB vaccine in HIV-infected, BCG-vaccinated adults with CD4(+) T cell counts >350 cells/mm(3). Vaccine. 2015 Apr 8;33(15):1890-6. doi: 10.1016/j.vaccine.2015.02.004. Epub 2015 Feb 17. PMID 25698492
- See also: Aurum Institute — http://www.auruminstitute.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo Control: Placebo was the identical buffer solution in which AERAS-402 is formulated.
Period: Overall Study
Arm/Group | Placebo | Investigational Vaccine
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Investigational Vaccine | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (6.49) | 30.5 (5.88) | 30.7 (6.07)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  South Africa | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: CD4+ Lymphocyte Count
Description: Assess the effect of AERAS-402 on the CD4+ lymphocyte count after 6 months in HIV-infected, BCG-vaccinated adult subjects with no evidence of active tuberculosis (TB disease) Change in cells/mm^3 pre-vaccination to Study Day 182
Time Frame: CD4+ counts from samples collected on Study days 0 and 182.
Measure: Median (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Placebo | Investigational Vaccine
Number analyzed (Participants) | 13 | 13
cells/mm^3 | -136.0 [-205.0 to 1.0] | -107.0 [-274.0 to -31.0]

2. Secondary Outcome: Change in HIV Viral Load in HIV-infected, BCG-vaccinated Adult Subjects Before and After Administration of AERAS-402 (From Day 1 to Day 182)
Time Frame: 6 months (day 182) post Study Day 0 vaccination.
Measure: Median (95% Confidence Interval); unit: Change in copies/mL over time
Arm/Group | Placebo | Investigational Vaccine
Number analyzed (Participants) | 13 | 13
Change in copies/mL over time | -0.163 [-0.274 to 0.336] | -0.011 [-0.357 to 0.281]

3. Secondary Outcome: Mtb-specific T Cell Response in HIV-infected BCG-vaccinated Adult Subjects With no Evidence of TB Disease
Description: Intracellular cytokine staining (ICS) assay immune response was expressed as the percentage of CD4+ and CD8+ T cells producing any one of three cytokines (IFN-γ, TNF-α, or IL-2) or any combination of the three cytokines simultaneously after stimulation with Ag85A, Ag85B, and TB10.4 peptide pools.
Time Frame: Study days 28 and 56
Population: percentage of CD4 or CD8 T-cell response
Measure: Median (95% Confidence Interval); unit: percentage of T-cell response
Arm/Group | Placebo | Investigational Vaccine
Number analyzed (Participants) | 13 | 13
percentage of T-cell response
  CD4+ Ag85A response at study day 28 | 0.0103 [0.0000 to 0.0230] | 0.0908 [0.0242 to 0.1357]
  CD4+ Ag85A response at study day 56 | 0.0199 [0.0000 to 0.0307] | 0.1248 [0.0537 to 0.2184]
  CD4+ Ag85B response at study day 28 | 0.0011 [0.0000 to 0.0166] | 0.0819 [0.0338 to 0.1069]
  CD4+ Ag85B response at study day 56 | 0.0083 [0.0000 to 0.0277] | 0.0769 [0.0426 to 0.1463]
  CD4+ TB10.4 response at study day 28 | 0.0196 [0.0027 to 0.0494] | 0.0364 [0.0133 to 0.0463]
  CD4+ TB10.4 response at study day 56 | 0.0281 [0.0070 to 0.0444] | 0.0443 [0.0223 to 0.1435]
  CD8+ Ag85A response at study day 28 | 0.0002 [0.0000 to 0.0019] | 0.0127 [0.0019 to 0.0462]
  CD8+ Ag85A response at study day 56 | 0.0027 [0.0000 to 0.0204] | 0.0300 [0.0040 to 0.0824]
  CD8+ Ag85B response at study day 28 | 0.0000 [0.0000 to 0.0100] | 0.0317 [0.0000 to 0.1140]
  CD8+ Ag85B response at study day 56 | 0.0040 [0.0000 to 0.0179] | 0.0846 [0.0113 to 0.1818]
  CD8+ TB10.4 response at study day 28 | 0.0000 [0.0000 to 0.0034] | 0.0000 [0.0000 to 0.0112]
  CD8+ TB10.4 response at study day 56 | 0.0051 [0.0000 to 0.0157] | 0.0094 [0.0000 to 0.0404]

ADVERSE EVENTS:
Description: Systematic Assessment of AEs by Diary Card, regular laboratory and investigator assessments. As well as subject-reported events.
Arm/Group | Placebo | Investigational Vaccine
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Investigational Vaccine (N=13)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Investigational Vaccine (N=13)
Acute sinusitis (Infections and infestations) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 5 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (5) | 4 (4)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (3)
Conjunctivitis (Eye disorders) | 2 (2) | 3 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 4 (11)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 6 (16)
Injection site erythema (General disorders) | 0 (0) | 4 (5)
Injection site induration (General disorders) | 0 (0) | 3 (4)
Injection site pain (General disorders) | 2 (2) | 10 (12)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 2 (2) | 5 (7)
Blood pressure systolic decreased (Investigations) | 3 (3) | 0 (0)
Blood pressure systolic increased (Investigations) | 3 (3) | 3 (3)
Blood urine present (Investigations) | 2 (2) | 4 (4)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Glucose urine (Investigations) | 0 (0) | 2 (3)
Haemoglobin decreased (Investigations) | 1 (1) | 4 (4)
Heart rate decreased (Investigations) | 0 (0) | 2 (3)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 5 (6)
Nitrite urine present (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Protein urine (Investigations) | 3 (3) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2)
White blood cells urine (Investigations) | 0 (0) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No